CLINICAL TRIAL: NCT01766336
Title: A 36-Week Safety Extension Study of Oral ELND005 for Treatment of Agitation and Aggression in Patients With Moderate to Severe Alzheimer's Disease
Brief Title: A 36-Week Safety Extension Study of ELND005 as a Treatment for Agitation and Aggression in Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELND005-AG251; 2012-005524-15 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease
Keywords: Agitation; Aggression; AD patients
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Aggression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 ELND005/ELND005 (Experimental): Patients who received ELND005 during Study AG201 will continue on the same maintenance dose for 36 weeks.
  Interventions: Drug: Group 1 ELND005
- Group 2 PLACEBO/ELND005 (Experimental): Patients who received placebo during Study AG201 will receive ELND005 at the same dosing regimen as the active group in Study AG201 for 36 weeks.
  Interventions: Drug: Group 2 ELND005

INTERVENTIONS:
Drug: Group 1 ELND005
  Arms: Group 1 ELND005/ELND005
Drug: Group 2 ELND005
  Arms: Group 2 PLACEBO/ELND005

SUMMARY:
To evaluate the safety and tolerability of ELND005 treatment with up to 36 weeks exposure, in Moderate to Severe AD patients with agitation and aggression.

ELIGIBILITY:
Inclusion Criteria:

* Complete Week 12 visit of AG201
* Both patient and study partner/caregiver are willing and able to participate in all scheduled evaluations and complete all required tests

Exclusion Criteria:

* Is currently using any other investigational or experimental drugs or devices
* Has significant worsening of medical conditions or dementia such that it may preclude completion of this safety extension study

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (38):
  - TransitionTIL Investigational Site, Birmingham, Alabama
  - TransitionTIL Investigational Site, Phoenix, Arizona
  - TransitionTIL Investigational Site, Encino, California
  - TransitionTIL Investigational Site, Escondido, California
  - TransitionTIL Investigational Site, Fresno, California
  - TransitionTIL Investigational Site, Long Beach, California
  - TransitionTIL Investigational Site, Newport Beach, California
  - TransitionTIL Investigational Site, Orange, California
  - TransitionTIL Investigational Site, Norwalk, Connecticut
  - TransitionTIL Investigational Site, Washington D.C., District of Columbia
  - TransitionTIL Investigational Site, Atlantis, Florida
  - TransitionTIL Investigational Site, Deerfield Beach, Florida
  - TransitionTIL Investigational Site, Delray Beach, Florida
  - TransitionTIL Investigational Site, Lake Worth, Florida
  - TransitionTIL Investigational Site, Oakland Park, Florida
  - TransitionTIL Investigational Site, Orlando, Florida
  - TransitionTIL Investigational Site, Port Charlotte, Florida
  - TransitionTIL Investigational Site, Sarasota, Florida
  - TransitionTIL Investigational Site, Columbus, Georgia
  - TransitionTIL Investigational Site, Savannah, Georgia
  - TransitionTIL Investigational Site, Springfield, Illinois
  - TransitionTIL Investigational Site, Easton, Maryland
  - TransitionTIL Investigational Site, Winchester, Massachusetts
  - TransitionTIL Investigational Site, Saint Paul, Minnesota
  - TransitionTIL Investigational Site, Rochester, New York
  - TransitionTIL Investigational Site, Charlotte, North Carolina
  - TransitionTIL Investigational Site, Durham, North Carolina
  - TransitionTIL Investigational Site, Wilmington, North Carolina
  - TransitionTIL Investigational Site, Winston-Salem, North Carolina
  - TransitionTIL Investigational Site, Oklahoma City, Oklahoma
  - TransitionTIL Investigational Site, Portland, Oregon
  - TransitionTIL Investigational Site, Abington, Pennsylvania
  - TransitionTIL Investigational Site, Jenkintown, Pennsylvania
  - TransitionTIL Investigational Site, Norristown, Pennsylvania
  - TransitionTIL Investigational Site, Pittsburgh, Pennsylvania
  - TransitionTIL Investigational Site, Port Royal, South Carolina
  - TransitionTIL Investigational Site, DeSoto, Texas
  - TransitionTIL Investigational Site, Bellevue, Washington
- TransitionTIL Investigational Site, Toronto, Ontario, Canada
- Spain (4):
  - TransitionTIL Investigational Site, Elche, Alicante
  - TransitionTIL Investigational Site, Terrassa, Barcelona
  - TransitionTIL Investigational Site, Barcelona
  - TransitionTIL Investigational Site, Madrid
- TransitionTIL Investigational Site, Swindon, Wiltshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- ELND005/ELND005: Patients who received ELND005 in AG201 and received ELND005 in this extension study AG251
- Placebo/ELND005: Patients who received Placebo in AG201 and received ELND005 in this extension study AG251
Period: Overall Study
Arm/Group | ELND005/ELND005 | Placebo/ELND005
Started | 150 | 146
Completed | 60 | 71
Not Completed | 90 | 75
Not completed — Adverse Event | 11 | 8
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor Decision | 52 | 43
Not completed — Withdrawal by Subject | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELND005/ELND005 | Placebo/ELND005 | Total
Number analyzed (Participants) | 150 | 146 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (7.9) | 75.9 (8.7) | 76.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 81 | 165
  Male | 66 | 65 | 131
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 2
  Black or African American | 10 | 17 | 27
  White | 138 | 127 | 265
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  North America | 137 | 134 | 271
  Europe | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events
Description: To evaluate the safety and tolerability of ELND005 treatment with up to 36 weeks exposure, in Moderate to Severe AD patients with agitation and aggression.
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | ELND005/ELND005 | Placebo/ELND005
Number analyzed (Participants) | 150 | 146
participants | 105 | 91

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient starting from the time the consent form was signed until the completion of the study.
Arm/Group | ELND005/ELND005 | Placebo/ELND005
Serious Adverse Events (participants affected / at risk) | 29/150 | 26/146
Other Adverse Events (participants affected / at risk) | 41/150 | 26/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELND005/ELND005 (N=150) | Placebo/ELND005 (N=146)
Syncope (Nervous system disorders) | 3 | 1
Dementia alzheimer's type (Nervous system disorders) | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Brain hypoxia (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Mental status change (Psychiatric disorders) | 3 | 3
Agitation (Psychiatric disorders) | 1 | 3
Aggression (Psychiatric disorders) | 1 | 0
Homocidial ideation (Psychiatric disorders) | 0 | 1
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
General physical health deterioriation (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELND005/ELND005 (N=150) | Placebo/ELND005 (N=146)
Agitation (Psychiatric disorders) | 15 | 14
Fall (Injury, poisoning and procedural complications) | 20 | 7
Urinary tract infection (Infections and infestations) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less